CLINICAL TRIAL: NCT01953146
Title: Timing of Development in Embryos Derived From Women With Polycystic Ovairan Syndrome and Controls
Brief Title: The Influence of Polycystic Ovairan Syndrome on Embryonic Developmental Timing
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Helene Nørrelund, Consultant, University of Aarhus
Other Study IDs: PCOS_time-lapse
Record Dates: First submitted 2013-09-23; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovarian Disease
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCOS criteria: nfertile patients undergoing assisted reproduction were consecutively recruited at the Fertility Clinic, Arhus University Hospital from February 2011 to May 2013. Women aged < 38 years without endometriosis where more than > 8 oocytes were retrieved were eligible. Patients were categorized in PCOS and non-PCOS according to the Rotterdam criteria for PCOS, defined by the presence of anovulation and polycystic ovaries.

SUMMARY:
Polycystic ovary syndrome is one of the most common causes of female infertility. The cause of infertility in PCOS is unknown. Factors other than anovulation, including inherited or induced changes in the embryo quality have been suggested. Time-lapse analysis of embryo development is a sensitive method of detecting reduced embryo viability. Yet, there are no data regarding the embryo development in PCOS assessed by time-lapse analysis.

DETAILED DESCRIPTION:
Method A consecutive cohort of 249 infertile women attending In vitro fertilization (IVF) or Intra-cytoplasmic sperm injection (ICSI) treatment at the Fertility Clinic, Arhus University Hospital was requited from February 2011 to May 2013. During the period, couples undergoing IVF/ICSI treatment were offered blastocyst culture to day 6 and time-lapse imaging (TLI) as part of a study evaluating parameters for embryo selection (Kirkegaard et al. 2013). Women aged < 38 years without endometriosis and with more than > 8 oocytes retrieved were eligible. Patients were categorized in two groups. Women with regular menstrual cycles and no clinical signs of PCOS (non-PCOS) and women fulfilling the Rotterdam diagnostic criteria for PCOS detected by the presence of anovulation and polycystic ovaries PCO, which was diagnosed by luteal-phase progesterone testing and trans-vaginal ultrasound, respectively. Biochemical parameters of androgen excess were included in the diagnosis when available, , whereas subjective symptoms of androgen excess (acne, hirsutism, alopecia) were not included.

Ethical approval Written informed consent was obtained from all patients before inclusion. The Central Denmark Region Committees on Biomedical Research Ethics and the Danish Data Protection Agency approved the study.

Ovarian stimulation:

Patients were treated with individual doses of gonadotropin, based on serum AMH and/or antral follicle count. Patients were stimulated by either a GnRH agonist- or antagonist protocol using rec-FSH or HMG for stimulation according to clinical guidelines. A dose of 10,000 IU of hCG was administered when at least 3 follicles measured ≥ 17 mm, and UL guided oocyte retrieval was conducted 36 h later.

Oocyte retrieval and ICSI/IVF Ovarian stimulation and oocyte retrieval were performed according to standard procedures. After fertilization, ICSI embryos were immediately placed in the time-lapse incubator (EmbryoScope™). IVF embryos were cultured for approximately 18 h in a conventional incubator. Before IVF embryos were transferred to the EmbryoScope, adhering cumulus cells were removed to ensure optimal image acquisition. In the EmbryoScope, all embryos were cultured until arrest or removal at day 6.

Embryo assessment. All embryos with 2 pronuclei completing the first cleavage were annotated manually.The following parameters were annotated with time-points: appearance and disappearance of 1st nucleus and 2nd nucleus after 1st division, 1st - 7th divisions, final divisions, compaction, morula, early and full expanded blastocyst, start of hatching and fully hatched blastocyst. All time-points were normalized to first cleavage and treated as durations for further analysis in order to overcome the limitation of inexact starting points, and facilitate comparison between IVF and ICSI populations. For the same reason, no parameters before first cleavage were investigated. Durations of cell cycles and cell stages were subsequently calculated as the interval between two time-points. Two parameters (multi-nucleation and direct cleavage to 3-cell stage) were assessed by binary values yes and no. Embryos were selected for transfer according to conventional measures of morphological quality on day 6 according to the Gardner criteria (Gardner et al. 2004) . No time-lapse parameters were used in the selection process. The observer was blinded to the patient's treatment data and medical history.

Statistics The influence of PCOS on embryo development was tested in regression models for clustered data. A covariance regression model was used to account for potential confounding variables: female age, BMI and fertility treatment. In total, 313 embryos from 43 PCOS women, and 1080 embryos from 175 non-PCOS women were analyzed.

ELIGIBILITY:
Inclusion Criteria:

Women aged < 38 years without endometriosis and with more than > 8 oocytes retrieved were eligible. -

Exclusion Criteria:

* All embryos with more or less than 2 pronuclei, and that did not undergo first cleavage were excluded

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A consecutive cohort of 249 infertile women attending In vitro fertilization (IVF) or Intra-cytoplasmic sperm injection (ICSI) treatment at the Fertility Clinic, Arhus University Hospital from February 2011 to May 2013.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Embryonic developmental timing assessed by Time-lapse analysis | From fertilization until transfer at day 6
  Embryos were cultured in a time-lapse incubator until arrest or removal at day 6. The time-point of an event was annotated and analyzed for the embryos in focus (in order of appearance).The influence of PCOS on embryo developmental timing was tested in regression models for patient-clustered data

CONTACTS AND LOCATIONS:
Overall Officials: Ulla B Knudsen, Professor, Study Director — Fertility Clinic Aarhus University
Locations (1):
- Fertility Clinic, Aarhus, N, Denmark

REFERENCES:
- [Derived] Sundvall L, Kirkegaard K, Ingerslev HJ, Knudsen UB. Unaltered timing of embryo development in women with polycystic ovarian syndrome (PCOS): a time-lapse study. J Assist Reprod Genet. 2015 Jul;32(7):1031-42. doi: 10.1007/s10815-015-0488-0. Epub 2015 May 1. PMID 25925351